CLINICAL TRIAL: NCT03281499
Title: A Pilot Study Integrating Transoral Robotic Surgery, Histopathologic Localization, and Tailored De-Intensification of Radiotherapy for Unknown Primary and Small Oropharyngeal Head and Neck Squamous Cell Carcinoma(FIND Trial)
Brief Title: Transoral Robotic Surgery and Tailored Radiotherapy in Unknown Primary and Small Squamous Cell Head and Neck Cancer
Acronym: FIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIND Trial
Record Dates: First submitted 2017-08-21; First posted 2017-09-13 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: There will only be a single group of participants in this study
Masking Description: No masking will be used in this study for both participants and the study team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- da Vinci Surgical System Model IS4000 (Experimental): Transoral robotic surgery, followed by tailored radiotherapy
  Interventions: Other: da Vinci Surgical System Model IS4000

INTERVENTIONS:
Other: da Vinci Surgical System Model IS4000 — tailored radiotherapy regimen following transoral robotic surgery
  Other Names: tailored radiotherapy regimen

SUMMARY:
The purpose of this study is to evaluate the use of Transoral Robotic Surgery (TORS) to identify small oropharyngeal carcinomas. Findings from this study will be used to better determine which patients may be suitable for more targeted radiotherapy that would lead to a reduction in the total amount of radiotherapy needed as part of their treatment. Reducing the amount of radiotherapy received has been found to reduce the risk of late complications and toxicity to the patient.The pathologic findings will then be used to determine patients who may be candidates for de-intensification of radiotherapy.

DETAILED DESCRIPTION:
Patients who present with carcinomas of unknown primary site (CUP) of the head and neck represent a challenging problem for clinicians both from a diagnostic and therapeutic perspective. Traditional techniques for identification of primary tumors involved a Positron Emission Tomography scan (PET)/ computerized tomography scan(CT) followed by examination under anesthesia with biopsies of the nasopharynx, tongue base, piriform sinuses in conjunction with a tonsillectomy may identify as many as 44% of primary tumors, the remaining unidentified tumors are treated with mucosal irradiation to all high risk mucosal sites. The addition of a lingual tonsillectomy with Transoral Robotic Surgery (TORS) may identify almost 70% of primary tumours that have otherwise escaped initial identification at this timepoint,. Historically, for those whose primary would not be discovered at the PET/CT, the discovery would have been made later during follow up visits.

The investigators propose to integrate Transoral Robotic Surgery into the diagnostic evaluation of participants presenting with metastatic squamous cell carcinoma to the neck of unknown primary origin. The investigators will localize small hidden oropharyngeal carcinomas, determine their laterality, and based on the laterality of the tumour, laterality of neck nodes, and completeness of resection, will offer reduced radiotherapy to the primary site and/or to the neck (de-intensification)to the participant. The investigators hypothesize that this approach to unknown primary carcinomas will be both safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Metastatic squamous cell carcinoma (T0,N1-3,M0) to at least one regional lymph node of the neck (includes N1-N3) based on fine needle aspiration (FNA) biopsy, core biopsy, excisional biopsy, or neck dissection
* Ability to understand and willing to sign a written informed consent document
* Women of child-producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication.

Exclusion Criteria:

* Evidence of a nasopharyngeal carcinoma by one or more of the following methods: endoscopic examination, imaging, positive nasopharyngeal biopsy or core lymph node biopsy staining for Epstein Barr Encoded RNA (EBER) by In Situ Hybridization.
* Prior non-cutaneous head and neck squamous cell carcinoma
* Prior head and neck radiotherapy
* History of neck dissection - contralateral to the side of the nodal disease
* Presence of lymphadenopathy on CT unlikely to originate from a primary oropharyngeal carcinoma (i.e., parotid, isolated low (level IV/low level V)
* Radiologically abnormal/enlarged retropharyngeal adenopathy.
* Poor performance status (ECOG status 3 - 5)
* Severe comorbidity or uncontrolled inter-current illness (i.e., unstable angina or heart failure in last 6 months, myocardial infarction in last 6 months, chronic obstructive pulmonary disease with exacerbations necessitating hospitalization or emergency room visit in the past 3 months, history of pneumonia in the past 3 months, use of home oxygen, uncorrectable coagulopathy)
* Not a surgical candidate
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Determination of the rate of out-of-field failures following treatment | 2 years
  The primary outcome for the study is to determine the rate of out-of-field failures following treatment as determined by use of morphologic imaging (contrast enhanced CT or MRI of the head) and confirmed by biopsy.

SECONDARY OUTCOMES:
Adverse Events (AE) monitoring | 2 years
  To determine the profile of TORS related complications and Surgical Adverse Events within 30 days of surgery using National Cancer Institute Common Terminology Criteria (CTC) for Adverse Events (NCI CTC-AE v 4.0)
Determination of proportions of occult oropharyngeal cancers identified | 2 years
  To determine the proportion of patients with occult oropharyngeal cancers identified
Location of primary tumours identified through enumeration of patients in each identified site group | 2 years
  To determine the location of primary tumours identified through enumeration of patients in each identified site group. The study data will be sorted by location of primary tumour and the proportions for each location calculated
Determination of the proportion of patients with completely resected primary tumours | 2 years
  To determine the location of primary tumours identified, the proportion of patients with primary oropharyngeal carcinomas completely resected (with negative margins), and the proportion of patients amenable to de-intensification treatment (ie, patients who receive no radiotherapy to the primary site and/or unilateral neck radiotherapy).
Determination of the proportion of patients patients amenable to de-intensification treatment | 2 years
  Determination of the proportion of patients patients amenable to de-intensification treatment
Exploration of expert rated swallowing impairment | 2 years
  To explore expert rated swallowing impairment on video fluoroscopic swallow studies (VFSS) using the Modified Barium Swallow Impairment (MBS-Imp)instrument tool 2 years
Exploration of patient reported swallowing related quality of life | 2 years
  To explore patient reported swallowing related quality of life using the MD Anderson Dysphagia Inventory (MDADI)
Exploration of speech and swallowing performance status | 2 years
  To explore observer rated speech and swallowing using the Performance Status Scale for Head and Neck (PSS-HN) instrument
Exploration of patient reported neck impairment | 2 years
  To explore patient reported neck impairment using the Neck Dissection Impairment Index (NDII) instrument
Determination of patterns of failure by location | 2 years
  To determine patterns of failure by location (local, regional, distant) as determined by CT/MRI of the Head and Neck and/or biopsy.
Rates of survival after treatment | 2 years
  To determine rates of survival at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John de Almeida, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kostakoglu L, Fardanesh R, Posner M, Som P, Rao S, Park E, Doucette J, Stein EG, Gupta V, Misiukiewicz K, Genden E. Early detection of recurrent disease by FDG-PET/CT leads to management changes in patients with squamous cell cancer of the head and neck. Oncologist. 2013;18(10):1108-17. doi: 10.1634/theoncologist.2013-0068. Epub 2013 Sep 13. PMID 24037978
- [Background] Strojan P, Ferlito A, Medina JE, Woolgar JA, Rinaldo A, Robbins KT, Fagan JJ, Mendenhall WM, Paleri V, Silver CE, Olsen KD, Corry J, Suarez C, Rodrigo JP, Langendijk JA, Devaney KO, Kowalski LP, Hartl DM, Haigentz M Jr, Werner JA, Pellitteri PK, de Bree R, Wolf GT, Takes RP, Genden EM, Hinni ML, Mondin V, Shaha AR, Barnes L. Contemporary management of lymph node metastases from an unknown primary to the neck: I. A review of diagnostic approaches. Head Neck. 2013 Jan;35(1):123-32. doi: 10.1002/hed.21898. Epub 2011 Oct 27. PMID 22034046
- [Background] Rodel RM, Matthias C, Blomeyer BD, Wolff HA, Jung K, Christiansen H. Impact of distant metastasis in patients with cervical lymph node metastases from cancer of an unknown primary site. Ann Otol Rhinol Laryngol. 2009 Sep;118(9):662-9. doi: 10.1177/000348940911800911. PMID 19810608
- [Background] Waltonen JD, Ozer E, Hall NC, Schuller DE, Agrawal A. Metastatic carcinoma of the neck of unknown primary origin: evolution and efficacy of the modern workup. Arch Otolaryngol Head Neck Surg. 2009 Oct;135(10):1024-9. doi: 10.1001/archoto.2009.145. PMID 19841343
- [Background] Jones AS, Cook JA, Phillips DE, Roland NR. Squamous carcinoma presenting as an enlarged cervical lymph node. Cancer. 1993 Sep 1;72(5):1756-61. doi: 10.1002/1097-0142(19930901)72:53.0.co;2-5. PMID 8348505
- [Background] Cianchetti M, Mancuso AA, Amdur RJ, Werning JW, Kirwan J, Morris CG, Mendenhall WM. Diagnostic evaluation of squamous cell carcinoma metastatic to cervical lymph nodes from an unknown head and neck primary site. Laryngoscope. 2009 Dec;119(12):2348-54. doi: 10.1002/lary.20638. PMID 19718744
- [Background] Chaturvedi AK, Anderson WF, Lortet-Tieulent J, Curado MP, Ferlay J, Franceschi S, Rosenberg PS, Bray F, Gillison ML. Worldwide trends in incidence rates for oral cavity and oropharyngeal cancers. J Clin Oncol. 2013 Dec 20;31(36):4550-9. doi: 10.1200/JCO.2013.50.3870. Epub 2013 Nov 18. PMID 24248688
- [Background] D'Souza G, Kreimer AR, Viscidi R, Pawlita M, Fakhry C, Koch WM, Westra WH, Gillison ML. Case-control study of human papillomavirus and oropharyngeal cancer. N Engl J Med. 2007 May 10;356(19):1944-56. doi: 10.1056/NEJMoa065497. PMID 17494927
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- [Background] Ali AN, Switchenko JM, Kim S, Kowalski J, El-Deiry MW, Beitler JJ. A model and nomogram to predict tumor site origin for squamous cell cancer confined to cervical lymph nodes. Cancer. 2014 Nov 15;120(22):3469-76. doi: 10.1002/cncr.28901. Epub 2014 Jul 24. PMID 25060659
- [Result] Abuzeid WM, Bradford CR, Divi V. Transoral robotic biopsy of the tongue base: A novel paradigm in the evaluation of unknown primary tumors of the head and neck. Head Neck. 2013 Apr;35(4):E126-30. doi: 10.1002/hed.21968. Epub 2011 Dec 16. PMID 22180229
- [Derived] de Almeida JR, Martino R, Hosni A, Goldstein DP, Bratman SV, Chepeha DB, Waldron JN, Weinreb I, Perez-Ordonez B, Yu E, Metser U, Hansen AR, Xu W, Su SJ, Kim J. Transoral Robotic Surgery and Radiation Volume Deintensification in Unknown Primary Squamous Cell Carcinoma of the Neck: The Phase 2 FIND Nonrandomized Controlled Trial. JAMA Otolaryngol Head Neck Surg. 2024 Jun 1;150(6):463-471. doi: 10.1001/jamaoto.2024.0423. PMID 38602692
- [Derived] de Almeida JR, Noel CW, Veigas M, Martino R, Chepeha DB, Bratman SV, Goldstein DP, Hansen AR, Yu E, Metser U, Weinreb I, Perez-Ordonez B, Xu W, Kim J. Finding/identifying primaries with neck disease (FIND) clinical trial protocol: a study integrating transoral robotic surgery, histopathological localisation and tailored deintensification of radiotherapy for unknown primary and small oropharyngeal head and neck squamous cell carcinoma. BMJ Open. 2019 Dec 30;9(12):e035431. doi: 10.1136/bmjopen-2019-035431. PMID 31892671